CLINICAL TRIAL: NCT05128188
Title: Sodium Accumulation Study In Haemodialysis
Brief Title: SASH: Sodium Accumulation Study In Haemodialysis
Acronym: SASH
Status: Completed | Type: Observational
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nicholas Selby, Professor of Nephrology, University Hospitals of Derby and Burton NHS Foundation Trust
Other Study IDs: UHDB/2021/020
Record Dates: First submitted 2021-11-05; First posted 2021-11-19 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Haemodialysis; End Stage Renal Disease on Dialysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients on haemodialysis: 5 patients on haemodialysis will be recruited. The study involves a single dialysis session and two MRI scans (one prior and one following dialysis) and collection of clinical data.
  Interventions: Other: No intervention will be given in this study

INTERVENTIONS:
Other: No intervention will be given in this study — No intervention will be given in this study

SUMMARY:
Haemodialysis (HD) sustains life in patients with end-stage kidney disease (ESKD) but is associated with a marked increase in incidence of cardiovascular disease (CVD) and high annual mortality rates. The pathogenesis of CVD in patients on HD is multifactorial and complex but hypertension is thought to be a major contributing factor. Sodium balance is normally regulated by the kidneys in health but has to be achieved by sodium removal during HD for those with ESKD. Recent evidence suggests that accumulation of sodium in the skin and / or muscle may be a critical factor impacting the development of hypertension and CVD in patients with ESKD and non-invasive methods are therefore required to study tissue sodium accumulation in this context. This study aims to determine the change in skin and muscle sodium content in patients undergoing haemodialysis. Participants will have a single haemodialysis session, and undergo two MRI scans (one prior to and one following dialysis).

DETAILED DESCRIPTION:
It has been proposed that tissue sodium accumulation in skin and/or muscle is a key factor in hypertension. 23Na MRI allows the assessment of skin and muscle sodium storage and will therefore be a valuable tool in elucidating the role of tissue sodium accumulation in the pathogenesis of salt-sensitive hypertension and cardiovascular morbidity and mortality. Moreover, if haemodialysis in patients with end-stage kidney disease (ESKD) results in changes in tissue sodium, the development of 23Na skin and muscle measures would allow for a method to correlate skin tissue sodium content with detailed cardiovascular and functional assessments.

Participants will have a single haemodialysis session, and undergo two MRI scans (one prior to and one following dialysis), in conjunction with clinical data collection (eg. blood samples, bioimpedance analysis, skin autoflorescence).

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years inclusive
* Male patients with CKD stage 5 receiving chronic haemodialysis
* Patient has been dialysis dependent for at least 3 months
* Must be able to follow simple instruction in English (on safety ground for MRI scans) and be able to understand the nature and requirements of the study

Exclusion Criteria:

* Active infection or malignancy
* Amputee
* Pregnancy
* Contraindication to MRI scanning including claustrophobia, pacemaker, metallic implants etc
* Unable or unwilling to provide informed consent
* Medical conditions or overall physical frailty precludes scan session in opinion of investigator
* Any condition which could interfere with the patient's ability to comply with the study

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 5 participants will be recruited from the renal unit
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Ascertainment of MRI measures of skin sodium content in 100% of patients studied | 6 months
  Sodium imaging of the skin and muscle of the upper calf will be performed using a range of sequences to quantify sodium in the skin and muscle using both fast-field-echo (FFE) and ultrashort TE (UTE) imaging techniques.
Ascertainment of MRI measures of muscle sodium content in 100% of patients studied | 6 months
  Sodium imaging of the skin and muscle of the upper calf will be performed using a range of sequences to quantify sodium in the skin and muscle using both fast-field-echo (FFE) and ultrashort TE (UTE) imaging techniques.

SECONDARY OUTCOMES:
To study skin sodium in haemodialysis patients and compare with previously reported healthy normal values | 6 months
  Sodium imaging of the skin and muscle of the upper calf will be performed using a range of sequences to quantify sodium in the skin and muscle using both fast-field-echo (FFE) and ultrashort TE (UTE) imaging techniques
To study muscle sodium in haemodialysis patients and compare with previously reported healthy normal values | 6 months
  Sodium imaging of the skin and muscle of the upper calf will be performed using a range of sequences to quantify sodium in the skin and muscle using both fast-field-echo (FFE) and ultrashort TE (UTE) imaging techniques
To measure degree of change in skin sodium content in relation to a single haemodialysis treatment | 6 months
  Quantification of sodium in skin and muscle and compare finding before and after dialysis
To measure degree of change in muscle sodium content in relation to a single haemodialysis treatment | 6 months
  Quantification of sodium in skin and muscle and compare finding before and after dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Selby, Professor, Principal Investigator — University Hospitals of Derby and Burton NHS Foundation Trust
Locations (1):
- University Hospitals of Derby and Burton NHS Foundation Trust, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No